CLINICAL TRIAL: NCT04824859
Title: A Geriatric Assessment Electronic Platform for Older Patients With Cancer (eGAP - Electronic Geriatric Assessment Platform)
Acronym: eGAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Technology issues
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Kah Poh Loh, Associate Professor - Department of Medicine, Hematology/Oncology (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCS21026
Record Dates: First submitted 2021-03-27; First posted 2021-04-01 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Cancer
Keywords: Supportive Care; Cancer; mHealth; Geriatric
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Electronic geriatric assessment platform to collect data (e.g., functional status, comorbidity, psychological health) that may better reflect health status of older adults with cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): The eGAP consists of validated questionnaires that are used to assess health status of older adults with cancer. Based on patient responses, tailored recommendations will be provided.
  Interventions: Behavioral: Behavioral

INTERVENTIONS:
Behavioral: Behavioral — eGAP that allows patients to complete validated questionnaires, and these questionnaires will be summarized and recommendations provided to the treating team

SUMMARY:
This project assesses the feasibility and usability of the geriatric assessment platform (electronic Geriatric Assessment Platform or eGAP in 50 older patients with cancer, their caregivers, and their oncology team. Using an iterative process, we will refine the eGAP based on input from stakeholders.

DETAILED DESCRIPTION:
A geriatric assessment is a multidisciplinary diagnostic process that can detect medical, psychosocial and functional problems not identified by routine evaluation. This can subsequently guide management of the identified problems. However, the time and resources required to incorporate a geriatric assessment into clinic visits remain the primary barriers for implementation. There is a need to increase the adoption of the geriatric assessment among general oncologists and to address the associated resource limitations. Our long-term goal is to utilize an electronic platform to facilitate completion of the geriatric assessment. This project assesses the feasibility and usability of the geriatric assessment platform (electronic Geriatric Assessment Platform or eGAP) in 50 older patients with cancer, their caregivers, and oncology providers. Using an iterative process, we will refine the eGAP based on input from stakeholders (patients, caregivers, oncologists, nurses, advanced practitioners)

ELIGIBILITY:
Inclusion Criteria for patients:

* Age ≥65 years
* Have a diagnosis of cancer
* Able to provide informed consent
* English-speaking (because the platform is currently in English)

Inclusion criteria for caregivers:

* Age ≥21 years
* Selected by patient when asked if there is a "family member, partner, friend, or caregiver with whom you discuss or who can be helpful in health-related matters".
* Able to provide informed consent
* English-speaking

Inclusion criteria for oncologists:

* Oncologists, APPs, and nurses who care for the patient

Exclusion Criteria:

* N/A

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility Retention Rate | 1 week
  Percentage of patients completing the assessments that are assigned to them on eGAP

SECONDARY OUTCOMES:
Recruitment rates | 1 week
  Percentage of patients who are approached and agree to enroll
Self-Report Completion Time | 1 week
  Time spent on completing the self-reported assessments on the eGAP
System Usability Scale | 1 week
  For patients, caregivers, and oncology providers: score on 10-item scale, ranging 0-100; higher score corresponds to greater usability

CONTACTS AND LOCATIONS:
Overall Officials: Kah Poh Loh, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A complete and final study protocol will be made publicly available through the University of Rochester Cancer Center Community Oncology Research Program Research Base Protocol and Data Sharing Committee. The full protocol and data will be made publicly available no later than the publication date of the study findings from the final dataset. The protocol will include a detailed description of the study population, hypotheses tested, measurement and assessment information, data definitions and codes, and the analysis plan utilized. We will be collecting identifying information. The final dataset will be stripped of identifiers prior to release for sharing. Published papers will be made available in portable document format.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available for 7 years from accrual of the first subject.